CLINICAL TRIAL: NCT01835457
Title: Concentration/Meditation as a Novel Means to Limit Inflammation: a Randomized Controlled Pilot Study
Brief Title: Concentration/Meditation Limits Inflammation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: LPS_concmed_controlled
Record Dates: First submitted 2013-03-25; First posted 2013-04-19 (Estimated); Last update posted 2013-07-23 (Estimated); Status verified 2013-03

CONDITIONS: Autoimmune Diseases
Keywords: Endotoxemia; Autonomic Nervous System; Inflammation; Meditation; Concentration; Iceman; LPS; Cortisol; Catecholamines
MeSH Terms: conditions — Autoimmune Diseases; Endotoxemia; Inflammation | interventions — Lipopolysaccharides; Meditation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Concentration/meditation group (Experimental): Subjects in this arm will be performing the concentration/meditation technique of Wim Hof (The Iceman) prior to, during and after intravenously injected 2 ng/kg Lipopolysaccharide
  Interventions: Drug: Lipopolysaccharide; Behavioral: Concentration/meditation
- Control group (Active Comparator): Subjects in this group will be intravenously injected with 2 ng/kg Lipopolysaccharide
  Interventions: Drug: Lipopolysaccharide

INTERVENTIONS:
Drug: Lipopolysaccharide — LPS is used to elicit an inflammatory response in all subjects.
  Other Names: Lipopolysaccharide (LPS) E. Coli 113:H 10:K negative
Behavioral: Concentration/meditation — A self-taught concentration/meditation technique that Mr Wim Hof developed himself, characterized by cycles consisting of a few minutes of hyperventilation followed by breath holding for up to 1-2 minutes and deep concentration (mindset).
  Other Names: Wim Hof Method
  Arms: Concentration/meditation group

SUMMARY:
Auto-immune diseases are characterized by an inappropriate inflammatory response against tissues in the body and represent a major health care burden. Pro-inflammatory cytokines such as TNF-α, IL-6 and IL-1β play a central role in the pathophysiology of many auto-immune diseases. Innovative therapies aimed at limiting pro-inflammatory cytokine production in a more physiological manner are warranted. In previous research conducted in an individual known as "the iceman", the investigators found that, through a autodidact concentration/meditation technique, he appears to mount a controlled stress response, characterized by activation of the sympathetic nervous system and enhanced production of cortisol, both of which are known to result in immunosuppression. In accordance, while practicing this concentration/meditation technique, the inflammatory response during human endotoxemia (lipopolysaccharide [LPS] administration) was remarkably low in this individual. Therefore, this technique could provide a novel means of controlling the inflammatory response. However, the aforementioned results were obtained in just one subject, and hence can not serve as scientific evidence for the effectiveness of the concentration/meditation technique. The iceman claims that he can teach this technique to other subjects within a relatively short time frame. Therefore, in the present study the investigators wish to investigate the effect of concentration/meditation on autonomic nervous system activity and the inflammatory response during experimental human endotoxemia in a controlled manner, by comparing a group of subjects that are trained by "the iceman" and practice the concentration/meditation technique with a group of subjects which do not.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 and ≤35 yrs
* Male
* Healthy
* Travel insurance (for travel to Poland for the training in the concentration/meditation technique)

Exclusion Criteria:

* Use of any medication
* Smoking
* Use of recreational drugs within 21 days prior to endotoxemia experiment day
* Use of caffeine or alcohol within 1 day prior to endotoxemia experiment day
* Previous participation in a trial where LPS was administered
* Surgery or trauma with significant blood loss or blood donation within 3 months prior to endotoxemia experiment day
* Participation in another clinical trial within 3 months prior to endotoxemia experiment day.
* History, signs, or symptoms of cardiovascular disease
* History of frequent vaso-vagal collapse or of orthostatic hypotension
* History of atrial or ventricular arrhythmia
* Hypertension (RR systolic >160 or RR diastolic >90)
* Hypotension (RR systolic <100 or RR diastolic <50)
* Conduction abnormalities on the ECG consisting of a 1st degree atrioventricular block or a complex bundle branch block
* Renal impairment: plasma creatinine >120 µmol/L
* Liver function abnormality: alkaline phosphatase>230 U/L and/or ALT>90 U/L
* History of asthma
* Obvious disease associated with immune deficiency.
* CRP > 20 mg/L, WBC > 12x109/L, or clinically significant acute illness, including infections, within 4 weeks before endotoxemia day

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-02; Primary Completion 2013-06 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Concentration of circulating TNF-α following LPS administration | 1 day

SECONDARY OUTCOMES:
Circulating cytokines (including but not limited to IL-6, IL-10 and IL1RA), following LPS administration. | 1 day
Body temperature after LPS administration | 1 day
Hemodynamic parameters after LPS administration | 1 day
  Blood pressure, heart rate, saturation, respiratory rate.
Plasma cortisol levels after LPS administration | 1 day
Plasma catecholamines levels after LPS administration | 1 day
Heart Rate Variability following LPS administration | 1 day
mtDNA concentrations following LPS administration | 1 day
Transcriptome analysis of circulating leukocytes after LPS administration | 1 day
Cytokine production by leukocytes ex vivo stimulated with LPS after LPS administration | 1 day
Changes in cell surface markers and functionality of circulating neutrophils after LPS administration | 1 day
effects of gut microbiome on inflammatory response elicited by LPS administration | 1 day
Ethylene and NO concentrations in exhaled breath after LPS administration | 1 day
Electrolyte concentrations in blood after concentration/meditation during endotoxemia | 1 day
Cortisol concentration in scalp hair | 1 measurement 3 weeks after LPS administration
Leukocyte counts and differentiation after LPS administration | 1 day
Illness symptoms after LPS administration | 1 day
  shivering, headache, back ache, muscle ache, vomiting.
Blood viscosity after LPS administration | 1 day
Platelet-leukocyte interactions after LPS administration | 1 day
  flow cytometric analysis of complexes between platelets on the one hand and monocytes, lymphocytes and neutrophils on the other hand.
beta-2 glycoprotein concentrations after LPS administration | 1 day
cell surface markers on circulating leukocytes after LPS administration | 1 day
Plasma endorphin levels after LPS administration | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: M. Kox, Dr., Principal Investigator — Intensive Care Medicine, Radboud University Nijmegen Medical Centre; P. Pickkers, MD, PhD, Study Director — Intensive Care Medicine, Radboud University Nijmegen Medical Centre
Locations (1):
- Intensive Care Medicine, Radboud University Nijmegen Medical Centre, Nijmegen, Gelderland, Netherlands